CLINICAL TRIAL: NCT06844253
Title: Comparative Effects of Exergaming Versus Task Oriented Training Among Sub-acute Post-stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/51
Record Dates: First submitted 2024-11-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Subacute Stroke
Keywords: Exergaming; Task-oriented training; Trunk control; sub-acute stroke; TIS; BBS
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Experimental): The participants will receive intervention through exergaming XBOX 360 which includes Kinect 20,000 leaks, Kinect bubble pop and Kinect rally ball trunk exercises.
  week 1-2 Kinect bubble pop (beginner level), Kinect 20000 leaks (beginner level) week 3-4 Kinect bubble pop (intermediate level), Kinect 20000 leaks (intermediate level) week5-6 Kinect rally ball (beginner level), Kinect bubble pop (advanced level) week7-8 Kinect rally ball (intermediate and advanced level) total 8 weeks. 3 days per week session will be given for 30 minutes including 5 minutes warm up and cool down and 5 minutes of break in between to avoid fatigue.
  Interventions: Procedure: INTERVENTION GROUP; TRAINING WITH EXERGAMING
- Control Group (Active Comparator): The participant will receive task oriented training consisting of different tasks in sitting and standing position.
  week1-2 sitting position: throwing and catching balls standing position: picking up glass from less heighted table . week 3-4 sitting position: transferring the plastic rings from one corner of table to another.
  standing position: catching balls from multiple directions. wee5-6 sitting position: picking objects from floor standing position: opening drawer from less heighted tables week 7-8 standing position: picking up and transferring bottles, jars at different locations on table standing position: removing stickers from wall time of session: 15-20 repetitions, 2 sets. 30 minutes of session with 5 minutes rest in between. the intervention will be given for 30 minutes , 3 days a week for total 8 weeks of time period.
  Interventions: Procedure: Task oriented training

INTERVENTIONS:
Procedure: INTERVENTION GROUP; TRAINING WITH EXERGAMING — RANDOMIZED CONTROL TRIAL EXERGAMING KINECT 20,000 LEAKS , KINECT BUBBLE POP, KINECT RALLY BALL GROUP 2: TASK ORIENTED TRAINING TRANSFERRING OBJECTS FROM ONE SIDE TO OTHER SIDE OF TABLE CATCHING AND THROWING BALLSIN DIFFERENT DIRECTIONS PICKING UP OBJECTS FROM LESS HIGHTED TABLES.
  Arms: Interventional Group
Procedure: Task oriented training — The participant will receive task oriented training consisting of different tasks in sitting and standing position.
  week1-2 sitting position: throwing and catching balls standing position: picking up glass from less heighted table . week 3-4 sitting position: transferring the plastic rings from one corner of table to another.
  standing position: catching balls from multiple directions. wee5-6 sitting position: picking objects from floor standing position: opening drawer from less heighted tables week 7-8 standing position: picking up and transferring bottles, jars at different locations on table standing position: removing stickers from wall time of session: 15-20 reps, 2 sets. 30 minutes of session with 5 minutes rest in between. the intervention will be given for 30 minutes , 3 days a week for total 8 weeks of time period.
  Arms: Control Group

SUMMARY:
This study is a randomized control trail and the purpose of this study is to determine the effects of exergaming versus task oriented training among sub-acute post-stroke patients.

DETAILED DESCRIPTION:
Effects of exergaming training will be assessed for trunk control which includes the parameters of balance and posture.

Sub-acute post stroke patients aged 40-85 years The participants will be assessed through Trunk impairment scale (TIS), Berg Blanace Scale (BBS) and biodex (clinical test for sensory integration in balance).

Informed consent will be taken after which the participants will be recruited into the two groups, where one group will receive intervention through exergaming and other group will receive task oriented trainig.

Baseline and post-treatment measurements will be taken for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sub-acute post-stroke.
* Aged 40 years-85 years.
* Mini-mental status examination >24
* Motor assessment scale (1-5 scoring)

Exclusion Criteria:

* Post-stroke patients with major cognitive deficits.
* Acute infections.
* Patients with any fracture/ MSK disorders.
* Neurological deficits other than stroke

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
TRUNK CONTROL | 8 weeks
  It will be assessed by trunk impairment scale. for trunk control : trunk impairment scale has total scoring 0-16. 0= severe impairment, 16=no impairment. trunk impairment scale will measure the trunk control in static sitting and static standing. and in rotational movements in left and right direction.
Balance | 8 weeks
  assessed by berg balance scale for balance berg balance scale has total scoring 56. 0-20=severe impairment, 21-40=moderate impairment, 41-56=mild impairment. berg balance scale will measure the static and dynamic balance in both sitting and standing position.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan